CLINICAL TRIAL: NCT04389177
Title: Efficacy and Safety of Pembrolizumab Plus Paclitaxel, Cisplatin Followed by Surgery in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma (KEYSTONE-001)
Brief Title: Pembrolizumab Plus Paclitaxel, Cisplatin Followed by Surgery for Locally Advanced ESCC (KEYSTONE-001)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TianjinCIH2020101
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2022-04

CONDITIONS: Esophageal Squamous Cell Carcinoma; Stage III
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — pembrolizumab; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab+ Paclitaxel+Cisplatin (Experimental): Pembrolizumab 200mg D1; Paclitaxel 135mg/m2 D2; Cisplatin 20mg/m2 D2-D4; repeated every 3 weeks
  Interventions: Drug: Pembrolizumab Injection [Keytruda]

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — Neoadjuvant period:preoperative therapy with three cycles: Pembrolizumab 200mg D1; Paclitaxel 135mg/m2 D2; Cisplatin 20mg/m2 D2-D4; repeated every 3 weeks.
  Da Vinci robot radical surgery: Before surgery, head/abdomen/chest CT scan, type B ultrasonic, upper gastrointestinal contrast, endoscopic ultrasound (EUS), and gastroscopy with biopsy will be done. Surgery should be done within 4-6 weeks after last neoadjuvant treatment finished.
  Adjuvant period: Adjuvant treatment with pembrolizumab 200mg every 3 weeks (6 cycles) should be performed within 3-6 weeks after surgery if the surgical pathology result is not pCR. abdomen/chest CT scan will be performed every 3 month after surgery.
  Other Names: Paclitaxel; Cisplatin

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of pembrolizumab plus paclitaxel, cisplatin followed by Da Vinci robot radical surgery for locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
The Preoperative chemoradiotherapy with surgery is the standard treatment in NCCN guideline. But many patients refused or abandon radiotherapy because of the intolerable adverse effects. We designed a single-arm, open-label, phase II trial of pembrolizumab plus paclitaxel, cisplatin followed by Da Vinci robot radical surgery for locally advanced (stage III) esophageal squamous cell cancer. The purpose of this study is to observe and evaluate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed esophageal squamous cell carcinoma;
2. Potentially resectable cT3N1M0，cT1-3N2M0(stage III)(AJCC 8 TNM classification);
3. Have a performance status of 0 or 1 on the ECOG Performance Scale;
4. Age 18-70 years old, both men and women;
5. Be willing and able to provide written informed consent/assent for the trial;
6. Demonstrate adequate organ function , all screening labs should be performed within 10 days of treatment initiation;
7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
8. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion through repeated biopsies. Newly-obtained is defined as a specimen obtained up to 4 weeks (28 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.

Exclusion Criteria:

1. Prior therapy (operation, radiotherapy, immunotherapy, or chemotherapy) for esophageal cancer;
2. Ineligibility or contraindication for esophagectomy;
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug;
4. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs);
5. Has severe hypersensitivity and adverse events (≥Grade 3) to nivolumab and/or any PD-1/PD-L1 inhibitors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | 3 months
  Viable tumor comprised ≤ 10% of resected tumor specimens

SECONDARY OUTCOMES:
Objective response rate (ORR) | 3 months
  Partial response is defined as a decrease by 30% or more in sums of longest diameter of measurable target lesions
Disease-free survival (DFS) | 24 months
  DFS is defined as the time interval between the date of enrollment and the date of the first documented evidence of relapse after radical resection at any site or death related to cancer (including toxicity), whichever occurred first.
Overall survival (OS) | 24 months
  Time from the enrollment to death of any cause
Lymph node derating rate | At time of surgery
  Lymph node derating rate
R0 resection rate | At time of surgery
  R0 resection rate

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobin Shang, MD,PhD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Department of minimally invasive esophageal surgery, Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shang X, Zhao G, Liang F, Zhang C, Zhang W, Liu L, Li R, Duan X, Ma Z, Yue J, Chen C, Meng B, Ren X, Jiang H. Safety and effectiveness of pembrolizumab combined with paclitaxel and cisplatin as neoadjuvant therapy followed by surgery for locally advanced resectable (stage III) esophageal squamous cell carcinoma: a study protocol for a prospective, single-arm, single-center, open-label, phase-II trial (Keystone-001). Ann Transl Med. 2022 Feb;10(4):229. doi: 10.21037/atm-22-513. PMID 35280363
- [Background] Lv H, Tian Y, Li J, Huang C, Sun B, Gai C, Li Z, Tian Z. Neoadjuvant Sintilimab Plus Chemotherapy in Resectable Locally Advanced Esophageal Squamous Cell Carcinoma. Front Oncol. 2022 Apr 29;12:864533. doi: 10.3389/fonc.2022.864533. eCollection 2022. PMID 35574384
- [Background] Shang X, Zhang W, Zhao G, Liang F, Zhang C, Yue J, Duan X, Ma Z, Chen C, Pang Q, Zhang W, Liu L, Ren X, Meng B, Zhang P, Ma Y, Zhang L, Li H, Kang X, Li Y, Jiang H. Pembrolizumab Combined With Neoadjuvant Chemotherapy Versus Neoadjuvant Chemoradiotherapy Followed by Surgery for Locally Advanced Oesophageal Squamous Cell Carcinoma: Protocol for a Multicentre, Prospective, Randomized-Controlled, Phase III Clinical Study (Keystone-002). Front Oncol. 2022 Mar 31;12:831345. doi: 10.3389/fonc.2022.831345. eCollection 2022. PMID 35433421
- [Background] Kassab J, Saba L, Kassab R, Kourie HR. Tsunami of immunotherapies in the management of esophageal cancer. Immunotherapy. 2022 Aug;14(11):879-884. doi: 10.2217/imt-2022-0035. Epub 2022 Jun 15. PMID 35703028
- [Background] Teixeira Farinha H, Digklia A, Schizas D, Demartines N, Schafer M, Mantziari S. Immunotherapy for Esophageal Cancer: State-of-the Art in 2021. Cancers (Basel). 2022 Jan 22;14(3):554. doi: 10.3390/cancers14030554. PMID 35158822
- See also: (Keystone-001): Interim analysis of a prospective, single-arm, single-center, phase II trial — http://doi.org/10.1016/j.annonc.2021.10.218